CLINICAL TRIAL: NCT02001558
Title: A Six Month Randomized Open-Label Trial of Pressure Ulcer Healing With Microcyn® Skin and Wound Care With Preservatives Versus Sterile Saline in Adult Spinal Cord Injury Subjects
Brief Title: Pressure Ulcer Healing With Microcyn
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Oculus Innovative Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Yu-ying Chen, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIC-UABWC-001
Record Dates: First submitted 2013-11-18; First posted 2013-12-05 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Pressure Ulcer; Spinal Cord Injuries
Keywords: Spinal cord injuries; Pressure ulcer
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries | interventions — Preservatives, Pharmaceutical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microcyn (Experimental): Microcyn is liberally sprayed on wound and permitted to remain on wound which will then be dressed with gauze that is moistened with Microcyn twice daily.
  Interventions: Drug: Microcyn
- Sterile saline (Active Comparator): Sterile saline is liberally sprayed on wound and permitted to remain on wound which will then be dressed with gauze that is moistened with sterile saline twice daily.
  Interventions: Other: Sterile saline

INTERVENTIONS:
Drug: Microcyn — Microcyn is liberally sprayed on wound and permitted to remain on wound which will then be dressed with gauze that is moistened with Microcyn twice daily for the earlier of total wound closure or Week 24
  Other Names: Microcyn® Skin and Wound Care with preservatives
  Arms: Microcyn
Other: Sterile saline — Sterile saline is liberally sprayed on wound and permitted to remain on wound which will then be dressed with gauze that is moistened with sterile saline twice daily for the earlier of total wound closure or Week 24
  Arms: Sterile saline

SUMMARY:
The purpose of this study is to test how well Microcyn™ works on Stage 3 and Stage 4 pressure ulcers compared to sterile saline among persons with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Persons with spinal cord injury
* Having Stage III/IV pressure ulcer(s)
* Able to fulfill all obligations of the study

Exclusion Criteria:

* Pressure ulcers scheduled for surgical closure within 14 days
* Use of any immunosuppressant medications within 30 days of screening
* Having conditions that put the subject at significant risk
* Medically unstable or has a life expectancy of less than 12 months
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Chen, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microcyn | Sterile Saline
Started | 32 | 33
Completed | 24 | 19
Not Completed | 8 | 14
Not completed — Lost to Follow-up | 8 | 14

BASELINE CHARACTERISTICS:
Population: Microcyn arm: there were 8 people were lost to follow up. Sterile saline arm: there were 14 people lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Microcyn | Sterile Saline | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.75 (13.37) | 39.24 (11.17) | 39.98 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 25 | 30 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 20 | 40
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at Baseline
Description: Pressure ulcer size is measured after debridement if debridement is provided. The pressure ulcer size (cubic centimeter) is the length (centimeter) times the width (centimeter) times the depth(centimeter). The range of value is from 0 to positive infinite.
Time Frame: pressure ulcer size (length x width x depth, cm^3) at baseline
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 32 | 33
cm^3 | 10.13 [0.38 to 196.00] | 21.00 [0.23 to 269.50]

2. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at 4 Weeks After Baseline
Description: as for outcome 1
Time Frame: 4 weeks after baseline
Population: Microcyn arm: there were 8 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 10 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 24 | 23
cm^3 | 9.00 [0.10 to 202.50] | 15.75 [0.00 to 160.00]

3. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at 8 Weeks After Baseline
Description: as for outcome 1
Time Frame: 8 weeks after baseline
Population: Microcyn arm: there were 12 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 17 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 20 | 16
cm^3 | 10.00 [0.23 to 216.13] | 20.06 [0.00 to 165.00]

4. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at 12 Weeks After Baseline
Description: as for outcome 1
Time Frame: 12 weeks after baseline
Population: Microcyn arm: there were 9 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 18 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 23 | 15
cm^3 | 7.50 [0.06 to 229.50] | 19.25 [0.00 to 224.00]

5. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at 16 Weeks After Baseline
Description: as for outcome 1
Time Frame: 16 weeks after baseline
Population: Microcyn arm: there were 13 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 19 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 19 | 14
cm^3 | 8.00 [0.01 to 267.75] | 11.63 [0.01 to 123.75]

6. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at 20 Weeks After Baseline
Description: as for outcome 1
Time Frame: 20 weeks after baseline
Population: Microcyn arm: there were 12 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 25 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 20 | 8
cm^3 | 7.63 [0.00 to 285.00] | 9.75 [0.00 to 72.00]

7. Primary Outcome: Pressure Ulcer Size (Length x Width x Depth, cm^3) at 24 Weeks After Baseline
Description: as for outcome 1
Time Frame: 24 weeks after baseline
Population: Microcyn arm: there were 12 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 19 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 20 | 14
cm^3 | 3.68 [0.05 to 200.00] | 8.68 [0.00 to 198.00]

8. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score
Description: PUSH categorizes pressure ulcer by surface area, exudate, and type of wound tissue. A comparison of total scores measured over time provides an indication of the improvement or deterioration in pressure ulcer healing. Total score ranges from 0 (healed, normal) to 17 (most severe).
Time Frame: at baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 32 | 33
score on a scale | 12.00 [4.00 to 15.00] | 12.00 [6.00 to 15.00]

9. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score at 4 Weeks After Baseline
Description: as for outcome 8
Time Frame: 4 weeks after baseline
Population: Microcyn arm: there were 8 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 12 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 24 | 21
score on a scale | 12.00 [5.00 to 17.00] | 11.00 [2.60 to 16.00]

10. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score at 8 Weeks After Baseline
Description: as for outcome 8
Time Frame: 8 weeks after baseline
Population: as for outcome 3
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 20 | 16
score on a scale | 11.00 [6.00 to 15.00] | 11.50 [0.00 to 15.00]

11. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score at 12 Weeks After Baseline
Description: as for outcome 8
Time Frame: 12 weeks after baseline
Population: Microcyn arm: there were 9 participants lost to follow up during this evaluation period.
  Sterile saline arm: there were 19 participants lost to follow up during this evaluation period.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 23 | 14
score on a scale | 10.00 [5.00 to 15.00] | 11.50 [0.00 to 15.00]

12. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score at 16 Weeks After Baseline
Description: as for outcome 8
Time Frame: 16 weeks after baseline
Population: as for outcome 5
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 19 | 14
score on a scale | 12.00 [2.00 to 14.00] | 11.50 [6.00 to 13.00]

13. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score at 20 Weeks After Baseline
Description: as for outcome 8
Time Frame: 20 weeks after baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 20 | 8
score on a scale | 11.00 [0.00 to 14.00] | 10.50 [0.00 to 14.00]

14. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score at 24 Weeks After Baseline
Description: as for outcome 8
Time Frame: 24 weeks after baseline
Population: as for outcome 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Microcyn | Sterile Saline
Number analyzed (Participants) | 20 | 14
score on a scale | 10.50 [4.00 to 15.00] | 11.00 [0.00 to 15.00]

ADVERSE EVENTS:
Time Frame: From baseline through 53 months.
Arm/Group | Microcyn | Sterile Saline
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT02001558/Prot_SAP_000.pdf